CLINICAL TRIAL: NCT06884111
Title: Single-Center, Randomized, Open, Exploratory, Drug Safety IIT Study of EE001 in Normal Adults/Patients with Mild, Moderate, or Severe (NYHA II-IV) Cardiac Insufficiency
Brief Title: Safety and Preliminary Efficacy Study of EE001 in Health/Patients Adults with Mild, Moderate, or Severe (NYHA II-IV) Cardiac Insufficiency
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui HygeianCells BioMedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHHCEE001CSP001
Record Dates: First submitted 2025-02-06; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-04

CONDITIONS: Cardiac Insufficiency
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: EE001，70-105ml per day by IV

INTERVENTIONS:
Drug: EE001，70-105ml per day by IV — EE001 is a brand-new testing agent for human studies, it is the first time in human being

SUMMARY:
This study is a single-center, randomized, open, exploratory, drug-safety IIT study of EE001 in normal adults/patients with mild, moderate, or severe (grades II-IV) cardiac insufficiency. Primary aims of this study is to assess the safety and tolerability of EE001 in normal adults and patients with mild, moderate, or severe (Class II-IV) cardiac insufficiency after single and consecutive repeated doses, and to carry out a preliminary evaluation of the pharmacodynamic indexes, to understand the preliminary efficacy of the drug in applied indications. The Secondary objectives are:

1. To observe the effect of EE001 on cardiac ejection index (color echocardiography) in normal adults and patients with mild, moderate or severe (Class II-IV) cardiac insufficiency;
2. To preliminarily evaluate the effect of EE001 on the cardiac functions of normal adults and patients with mild, moderate or severe (Class II-IV) cardiac insufficiency, in accordance with the comprehensive criteria of cardiac function index.
3. Six-minute walk test: to preliminarily assess the effect of EE001 on the exercise status of normal adults and patients with mild, moderate or severe (Class II-IV) cardiac insufficiency;
4. to assess the effect of EE001 on the serum levels of BNP and cardiac enzyme profiles of subjects after administration of EE001 to normal adults and patients with mild, moderate or severe (Class II-IV) cardiac insufficiency;
5. to evaluate the effect of EE001 on changes in human cytokine levels (IL-1, IL-6, IL-10, TNF-α, etc.) in normal adults and patients with mild, moderate or severe (Class II-IV) cardiac insufficiency; and
6. to evaluate the effect of EE001 on changes in the number of regulatory T cells in normal adults and patients with mild, moderate or severe (Class II-IV) cardiac insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1) Male and female subjects between 18 and 75 years of age (including upper and lower limits).

(2) Body Mass Index (BMI) between 19 and 28 kg/m2 (including upper and lower limits).

(3) Sperm and egg donation is prohibited during the study period (from signing of the Informed Consent Form to the final follow-up visit) and within 90 days of the final dose of study medication, and there is no likelihood of conception (or impregnation of a sexual partner), childbearing, or breastfeeding.

(4) No history of major medical problems, and there are no medical conditions during the screening period that may have contributed to the study.

no history of major diseases, and the results of physical examination, vital signs and laboratory tests during the screening period are normal, or out of the normal reference range but not clinically significant in the judgment of the investigator.

(5) The ability to communicate with clinical staff and comply with the requirements of the study.

(6) Signing the informed consent form to indicate their willingness to participate in the study.

Exclusion Criteria:

1. The presence of a medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the drug or that may interfere with adherence to the study protocol.
2. Have history of hemophilia or coagulation disorders.
3. Diagnosed with of endocrine, neurological, hematological, immunological (including hereditary immune deficiencies by personal or family history), psychiatric, metabolic abnormalities, lymphoproliferative disorders, severe or opportunistic infections (including herpes, tuberculosis) that in the opinion of the investigator are still clinically significant.
4. Allergies, particularly to eggs or chicken.
5. Participation in other clinical studies within 90 days prior to the first application of the investigational product.
6. Discontinuation of other, what in the opinion of the investigator, affects the results of the evaluation of this study, prior to the first application of the investigational product prescription or over-the-counter medication for less than 14 days or 5 half-lives of that medication (whichever is longer).
7. With history of malignancy within the past 5 years.
8. Having donated blood or lost a significant amount of blood (>400 mL) within 90 days prior to the first use of the investigational product.
9. Having undergone major surgery (as determined by the investigator based on past medical history information) or having suffered major trauma.
10. Subjects with abnormal vital sign measurements that are clinically significant in the judgment of the investigator.
11. Clinical or laboratory evidence of the presence of one of the following: Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), Human Immunodeficiency Virus (HIV), or syphilis carriage/infection.
12. With severe renal disease.
13. Difficulty with intravenous blood collection or known history of multiple episodes of needle or blood sickness.
14. Have history of regular alcohol consumption in the 6 months prior to screening, more than 14 drinks/week (1 drink = 5 oz wine or 12 oz beer or 1.5 oz spirits) in males, or exceeding the alcohol test limit during the Screening Period; who have taken any alcohol-containing product within 48 hours prior to the first use of the investigational product or who do not agree to avoid any alcohol-containing product during the trial period;
15. Poor compliance and unwillingness to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Safety assessment | Baseline, Day 1, Day7
  General toxicities and safe pharmacology properties of EE001 to human body at the applied dosage procedure will be assessed at different time point.

SECONDARY OUTCOMES:
Efficacy assessment | Baseline, Day1, Day7
  The preliminary efficacy of EE001 on cardiac ejection index (color echocardiography) at the applied administration schedule will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- AnHui Hygeiancells BioMedical Co., Ltd., Huangshan City, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes